CLINICAL TRIAL: NCT02591472
Title: An Integrated-Delivery-of-Care Approach to Improve Patient Outcomes, Safety, Well-Being After Orthopaedic Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Athletic Trainers' Association Research & Education Foundation (NATA Foundation) (Other); Foundation for Physical Medicine and Rehabilitation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201500753
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Musculoskeletal Injury Trauma
MeSH Terms: interventions — Delivery of Health Care, Integrated; Muscle Strength Dynamometer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (UsCare) (Active Comparator): This group will receive UsCare for orthopedic trauma involves surgical intervention, acute care therapies, post-acute rehabilitation and follow-up clinic visits after discharge. Additionally, the following test will be performed: Lower Extremity Gain Scale (LEGS), dynamometer isometric handgrip strength, Active Range of Motion (AROM), Posttraumatic Stress Disorder (PTSD), Beck Depression Inventory-II, State-Trait Anxiety Inventory (STAI), Tampa Scale of Kinesiophobia-11 (TSK-11), and Patient-Reported Outcomes Measurement Information System (PROMIS).
  Interventions: Procedure: Usual Care (UsCare); Other: Patient-Reported Outcomes Measurement Information System; Other: Lower Extremity Gain Scale (LEGS); Other: Dynamometer; Other: Active Range of Motion (AROM); Other: Posttraumatic Stress Disorder (PTSD); Other: Beck Depression Inventory-II; Other: State-Trait Anxiety Inventory (STAI); Other: Tampa Scale of Kinesiophobia-11 (TSK-11)
- Integrated Care (ICare) (Experimental): This group will receive ICare for orthopedic trauma involves surgical intervention, acute care therapies, post-acute rehabilitation and follow-up clinic visits after discharge, plus simultaneous psychosocial support via the Transform-10 Program.. Additionally, the following test will be performed: Lower Extremity Gain Scale (LEGS), dynamometer isometric handgrip strength, Active Range of Motion (AROM), Posttraumatic Stress Disorder (PTSD), Beck Depression Inventory-II, State-Trait Anxiety Inventory (STAI), Tampa Scale of Kinesiophobia-11 (TSK-11), and Patient-Reported Outcomes Measurement Information System (PROMIS).
  Interventions: Procedure: Integrated care (ICare); Other: Patient-Reported Outcomes Measurement Information System; Other: Lower Extremity Gain Scale (LEGS); Other: Dynamometer; Other: Active Range of Motion (AROM); Other: Posttraumatic Stress Disorder (PTSD); Other: Beck Depression Inventory-II; Other: State-Trait Anxiety Inventory (STAI); Other: Tampa Scale of Kinesiophobia-11 (TSK-11)

INTERVENTIONS:
Procedure: Integrated care (ICare) — The Integrated Care approach provides Usual Care processes plus simultaneous psychosocial support via the Transform-10 Program. The Transform-10 Program will include information regarding emotional well-being, social support, and provides opportunity for the patient to openly discuss their thoughts and concerns regarding their recovery. The patient's normal clinical care usually includes a hospital stay, a 2 week follow up, 6 week follow up, 12 week follow up, 6 month, and 1 year follow up visit.
  Other Names: ICare
  Arms: Integrated Care (ICare)
Procedure: Usual Care (UsCare) — Usual Care includes radiographic imaging and administration of pain medication and antibiotics, skin care and range of motion of the injured area. The patient's normal clinical care usually includes a hospital stay, a 2 week follow up, 6 week follow up, 12 week follow up, 6 month, and 1 year follow up visit. At the end of the study all of the materials that make up the Transform-10 Program will be provided.
  Other Names: UsCare
  Arms: Usual Care (UsCare)
Other: Patient-Reported Outcomes Measurement Information System — Questionnaires of Physical Functional quality of life and Emotional Well-being will be performed during the hospital stay, a 2 week follow up, 6 week follow up, 12 week follow up, 6 month, and 1 year follow up visit.
  Other Names: PROMIS
Other: Lower Extremity Gain Scale (LEGS) — LEGS consists of a 3-meter walk, putting on a sock, putting on a shoe, rising from an armless chair, stepping up and down stairs, getting on and off the toilet, reaching from a sitting position to an object on the ground. In people with traumatic fractures, LEGS has high internal consistency and the content, concurrent and construct validity are high. This assessment will be performed during the hospital stay, at the 2 week follow up, 6 week follow up, 12 week follow up, 6 month, and 1 year follow up visit.
Other: Dynamometer — Isometric handgrip strength will be measured using a hand-held hydraulic dynamometer. Handgrip strength is clinically important as it strongly predicts long-term function capability after orthopedic trauma. This assessment will be performed during the hospital stay, at the 2 week follow up, 6 week follow up, 12 week follow up, 6 month, and 1 year follow up visit.
  Other Names: Isometric handgrip strength
Other: Active Range of Motion (AROM) — The use of goniometer and a digital inclinometer will be used to assess AROM. This assessment will be performed during the hospital stay, at the 2 week follow up, 6 week follow up, 12 week follow up, 6 month, and 1 year follow up visit.
Other: Posttraumatic Stress Disorder (PTSD) — The Posttraumatic Stress Disorder (PTSD) Checklist will be administered to measure posttraumatic stress levels. This assessment will be performed during the hospital stay, at the 2 week follow up, 6 week follow up, 12 week follow up, 6 month, and 1 year follow up visit.
Other: Beck Depression Inventory-II — The Beck Depression Inventory-II is a broadly-applicable, clinically relevant psychometric instrument with high reliability and consistency which notes depression. This assessment will be performed during the hospital stay, at the 2 week follow up, 6 week follow up, 12 week follow up, 6 month, and 1 year follow up visit.
  Other Names: BDI-II
Other: State-Trait Anxiety Inventory (STAI) — The State-Trait Anxiety Inventory (STAI) will be used to measure state anxiety (anxiety about an event) and trait anxiety (anxiety level as a personal characteristic). This assessment will be performed during the hospital stay, at the 2 week follow up, 6 week follow up, 12 week follow up, 6 month, and 1 year follow up visit.
Other: Tampa Scale of Kinesiophobia-11 (TSK-11) — Tampa Scale of Kinesiophobia-11 (TSK-11) will be used to assess pain-related fear in orthopaedic trauma. This assessment will be performed during the hospital stay, at the 2 week follow up, 6 week follow up, 12 week follow up, 6 month, and 1 year follow up visit.

SUMMARY:
Orthopedic trauma is an unforeseen life-changing event. Nearly 2.8 million Americans sustain traumatic orthopedic injuries such as major fractures or amputation each year. Injury is treated in the hospital by physicians who medically stabilize and reconstruct the patient. Upon completion of their hospital stay, patients are discharged to begin their reintegration back into home and community activities. Despite high surgical success and survivorship rates, these injuries often result in poor quality of life (QOL)-related outcomes in otherwise healthy people. Fifty to ninety percent of patients develop severe psychological distress such as post-traumatic stress syndrome, depression or anxiety. Patients are often not provided the comprehensive support care and resources that are necessary to cope successfully with psychological stress and reintegrate into purposeful living. This is a major problem because high distress levels predict poor physical function, use of pain medications and low QOL. Survivors often cannot return to work, have persistent pain and experience social isolation. Distress worsens the self-perceptions of functional gain and efficacy and decreases personal fulfillment. Lingering psychological distress contributes to the development of other health problems and rebuilding of life is negatively impacted. The lack of psychosocial support contributes to injury re-occurrence, injury recidivism, re-hospitalizations and longer hospitalization stays, and higher personal and societal health care costs.

There is currently a lack of comparative efficacy research to determine which delivery approach produces greater improvements in the outcomes that are most desired by patients, specifically, functional QOL and emotional well-being. The proposed research will directly compare these delivery-of-care approaches and measure the patient-reported outcomes that are considered important to patients.

DETAILED DESCRIPTION:
The research study will determine whether the Usual Care or Integrated Care (which is Usual Care plus emotional support, and education/information during the hospital stay) helps patients feel better about their physical function and emotional well-being.

Participants with serious musculoskeletal injury, being treated at to the University of Florida's (UF) Orthopaedic Trauma service at UF Health at Shands Hospital, will be randomized (like tossing a coin) between the two groups.

Usual Care will follow all the highest standards for injury treatment.

Integrated Care will include medical care and emotional support. Study Staff are trained to provide emotional support and teach patients the skills for goal setting, taking ownership of journey, establishing lifelines, mobilizing resources and reducing stressors.

In addition, questionnaires and simple functional tests will be collected at the hospital and at normal follow-up visits at weeks 2, 6 and 12 and months 6 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with severe or multiple orthopedic trauma
* Patients who have received or will receive ≥1 surgical procedure for their orthopedic injuries
* Any major bone fractures that impairs mobility and/or participation in activities of daily living and self-care

Exclusion Criteria:

* Patients with a traumatic brain injury
* Patients with the inability to communicate effectively (e.g., at a level where self-report measures could be answered completely; such as medicated state or mechanically ventilated)
* Patients currently using psychotropic medications
* Patients with psychotic, suicidal or homicidal ideations.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-01-11; Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MaryBeth Horodyski, Ph.D., Principal Investigator — University of Florida Department of Orthopaedics
Locations (1):
- UF and Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States

REFERENCES:
- [Background] Castillo RC, Wegener ST, Newell MZ, Carlini AR, Bradford AN, Heins SE, Wysocki E, Pollak AN, Teter H, Mackenzie EJ. Improving outcomes at Level I trauma centers: an early evaluation of the Trauma Survivors Network. J Trauma Acute Care Surg. 2013 Jun;74(6):1534-40. doi: 10.1097/TA.0b013e3182921606. PMID 23694884
- [Background] Vincent HK, Horodyski M, Vincent KR, Brisbane ST, Sadasivan KK. Psychological Distress After Orthopedic Trauma: Prevalence in Patients and Implications for Rehabilitation. PM R. 2015 Sep;7(9):978-989. doi: 10.1016/j.pmrj.2015.03.007. Epub 2015 Mar 12. PMID 25772720
- [Background] Becher S, Smith M, Ziran B. Orthopaedic trauma patients and depression: a prospective cohort. J Orthop Trauma. 2014 Oct;28(10):e242-6. doi: 10.1097/BOT.0000000000000128. PMID 24736695
- [Background] Vranceanu AM, Bachoura A, Weening A, Vrahas M, Smith RM, Ring D. Psychological factors predict disability and pain intensity after skeletal trauma. J Bone Joint Surg Am. 2014 Feb 5;96(3):e20. doi: 10.2106/JBJS.L.00479. PMID 24500592
- [Background] Holbrook TL, Anderson JP, Sieber WJ, Browner D, Hoyt DB. Outcome after major trauma: 12-month and 18-month follow-up results from the Trauma Recovery Project. J Trauma. 1999 May;46(5):765-71; discussion 771-3. doi: 10.1097/00005373-199905000-00003. PMID 10338392
- [Background] Calder A, Badcoe A, Harms L. Broken bodies, healing spirits: road trauma survivor's perceptions of pastoral care during inpatient orthopaedic rehabilitation. Disabil Rehabil. 2011;33(15-16):1358-66. doi: 10.3109/09638288.2010.532280. Epub 2010 Nov 20. PMID 21091044
- [Background] Ponzer S, Molin U, Johansson SE, Bergman B, Tornkvist H. Psychosocial support in rehabilitation after orthopedic injuries. J Trauma. 2000 Feb;48(2):273-9. doi: 10.1097/00005373-200002000-00013. PMID 10697086
- [Derived] Zdziarski-Horodyski L, Horodyski M, Sadasivan KK, Hagen J, Vasilopoulos T, Patrick M, Guenther R, Vincent HK. An integrated-delivery-of-care approach to improve patient reported physical function and mental wellbeing after orthopedic trauma: study protocol for a randomized controlled trial. Trials. 2018 Jan 11;19(1):32. doi: 10.1186/s13063-017-2430-5. PMID 29325583

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care (UsCare): This group will receive UsCare for orthopedic trauma involves surgical intervention, acute care therapies, post-acute rehabilitation and follow-up clinic visits.
  Usual Care (UsCare) includes radiographic imaging and administration of pain medication and antibiotics, skin care and range of motion of the injured area. Normal clinical care usually includes a hospital stay, a 2 week, 6 week, and 12 week follow up visits. At the end of the study the materials for the Transform-10 Program will be provided. Additionally, the following tests will be performed:
  Patient-Reported Outcomes Measurement Information System: Questionnaires of Physical Functional quality of life and Emotional Well-being will be done during the 2 week, 6 week,12 week follow up visits.
  Lower Extremity Gain Scale (LEGS) consists of a 3-meter walk, putting on sock, putting on shoe, rising from a chair, stepping up/ down stairs, getting on/off the toilet, reaching from a sitting position to an object on the ground. This will be performed at the 6 week and 12 week follow up visits.
  Dynamometer: Isometric handgrip strength will be measured with a hand-held hydraulic dynamometer. This test will be performed at the 2 week, 6 week and 12 week follow up visits.
  Tampa Scale of Kinesiophobia-11 (TSK-11) will be used to assess pain-related fear in orthopaedic trauma. This will be performed at the 2 week, 6 week and 12 week follow up visits.
- Integrated Care (ICare): This group will receive ICare for orthopedic trauma involves surgical intervention, acute therapies, post-acute rehabilitation and follow-up clinic visits and simultaneous psychosocial support via the Transform-10 Program.
  Integrated care (ICare):This approach provides Usual Care plus the Transform-10 Program that includes information for emotional well-being, social support and opportunity for the patient to discuss thoughts and concerns with recovery. Patient's normal clinical care usually includes a hospital stay, a 2 week, 6 week, and 12 week follow up visits.
  Additionally, the following test will be performed:
  Patient-Reported Outcomes Measurement Information System: Questionnaires of Physical Functional quality of life and Emotional Well-being will be done during the 2 week, 6 week,12 week follow up visits.
  Lower Extremity Gain Scale (LEGS) consists of a 3-meter walk, putting on sock, putting on shoe, rising from a chair, stepping up/ down stairs, getting on/off the toilet, reaching from a sitting position to an object on the ground. This will be performed at the 6 week and 12 week follow up visits.
  Dynamometer: Isometric handgrip strength will be measured with a hand-held hydraulic dynamometer. This test will be performed at the 2 week, 6 week and 12 week follow up visits.
  Tampa Scale of Kinesiophobia-11 (TSK-11) will be used to assess pain-related fear in orthopaedic trauma. This will be performed at the 2 week, 6 week and 12 week follow up visits.
Period: Overall Study
Arm/Group | Usual Care (UsCare) | Integrated Care (ICare)
Started | 50 | 38
Completed | 50 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care (UsCare) | Integrated Care (ICare) | Total
Number analyzed (Participants) | 50 | 38 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 35 | 83
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (15.3) | 41.25 (18.1) | 42.23 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 33 | 21 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 5 | 14
  White | 31 | 32 | 63
  More than one race | 8 | 0 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 38 | 88

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline, at Weeks 2, 6 and 12 on the Patient Reported Outcome Measurement Information System (PROMIS) - Physical Function Between the Groups.
Description: Survey questionnaire measures the perception of Physical Function. Physical Function Average: t score = 50±10 Min: 10 Max: 90 A higher PROMIS T-score represents more of the concept being measured. For positively-worded concepts like Physical Functional T-score of 60 is one SD better than average. By comparison, a Physical Function T-score of 40 is one SD worse than average.
Time Frame: Change from baseline at weeks 2, 6 and 12
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Usual Care (UsCare) | Integrated Care (ICare)
Number analyzed (Participants) | 50 | 38
percentage of change from baseline
  2 weeks | 18.65 (26) | 17.6 (31.9)
  6 weeks | 25.8 (28.3) | 30.45 (33.05)
  12 weeks | 47.65 (37.9) | 41.35 (31.1)

2. Secondary Outcome: Change From Baseline at Weeks 6 and 12 on the Lower Extremity Gain Scale (LEGS) Between the Groups.
Description: LEGS consists combined score taken of a 3-meter walk, putting on a sock, putting on a shoe, rising from an armless chair, stepping up and down stairs, getting on and off the toilet, reaching from a sitting position to an object on the ground.
  Best score 27 Minimum score 0 Normal scores not available
Time Frame: Change from baseline at weeks 6 and 12
Measure: Mean (Standard Deviation); unit: percentage of change in LEGS score
Arm/Group | Usual Care (UsCare) | Integrated Care (ICare)
Number analyzed (Participants) | 50 | 38
percentage of change in LEGS score
  week 6 | 34.55 (35.55) | 46.8 (54.15)
  week 12 | 87.6 (66.45) | 232.25 (267.35)

3. Secondary Outcome: Change From Baseline at Weeks 2, 6 and 12 on the Tampa Scale of Kinesiophobia-11 (TSK-11) Between the Groups.
Description: Survey questionnaire given assess the pain-related fear of movement in orthopaedic trauma and the Tampa Scale of Kinesiophobia-11 (TSK-11) will be used. Best Score: 11 Min: 11 Max: 44
Time Frame: Change from baseline at weeks 2, 6 and 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UsCare) | Integrated Care (ICare)
Number analyzed (Participants) | 50 | 38
score on a scale
  week 2 | 26.1 (7.45) | 26.65 (5.37)
  week 6 | 24.5 (6.69) | 25 (6.48)
  week 12 | 23.15 (6.19) | 26 (7.45)

4. Secondary Outcome: Absolute Hand Grip Scores at Weeks 2, 6 and 12 on the Hand-held Hydraulic Dynamometer to Measure Handgrip Strength Between the Groups.
Description: Isometric handgrip strength is a valid predictor of mobility and will be measured using a hand-held hydraulic dynamometer.
  Average: 39 kg Range: 33-45 kg This is an estimated range for normal healthy subject. However, some of the patients in this study did not fall within this estimated range.
  The Unit of Measure is kilograms (kg). Subsequently all values presented are in kilograms (kg).
Time Frame: Absolute hand grip scores at weeks 2, 6 and 12
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Usual Care (UsCare) | Integrated Care (ICare)
Number analyzed (Participants) | 50 | 38
kilograms
  2 weeks | 31.35 (16.6) | 30.1 (19.15)
  6 weeks | 35.3 (15.8) | 30.9 (13.1)
  12 weeks | 35.9 (15.45) | 33.95 (12.8)

ADVERSE EVENTS:
Time Frame: From moment of consent until completion of study at 12 weeks.
Groups:
- Usual Care (UsCare): This group will receive UsCare for orthopedic trauma involves surgical intervention, acute care therapies, post-acute rehabilitation and follow-up clinic visits.
  Usual Care (UsCare) includes radiographic imaging and administration of pain medication and antibiotics, skin care and range of motion of the injured area. Normal clinical care usually includes a hospital stay, a 2 week, 6 week, and 12 week follow up visits. At the end of the study the materials for the Transform-10 Program will be provided. Additionally, the following tests will be performed:
  Patient-Reported Outcomes Measurement Information System: Questionnaires of Physical Functional quality of life and Emotional Well-being will be done during the 2 week, 6 week,12 week follow up visits.
  Lower Extremity Gain Scale (LEGS) consists of a 3-meter walk, putting on sock, putting on shoe, rising from a chair, stepping up/ down stairs, getting on/off the toilet, reaching from a sitting position to an object on the ground. This will be performed at the 6 week and 12 week follow up visits.
  Dynamometer: Isometric handgrip strength will be measured with a hand-held hydraulic dynamometer. This test will be performed at the 2 week, 6 week and 12 week follow up visits.
  Tampa Scale of Kinesiophobia-11 (TSK-11) will be used to assess pain-related fear in orthopaedic trauma. This will be performed at the 2 week, 6 week and 12 week follow up visits.ment
Arm/Group | Usual Care (UsCare) | Integrated Care (ICare)
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/38
Other Adverse Events (participants affected / at risk) | 0/50 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/72/NCT02591472/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT02591472/SAP_001.pdf